CLINICAL TRIAL: NCT01646528
Title: The Value of Mesenchymal Black Spots in Diagnosing Gastric Intestinal Metaplasia by Confocal Laser Endomicroscopy
Brief Title: The Value of Black Spots in Diagnosing Gastric Intestinal Metaplasia by Confocal Laser Endomicroscopy
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Shandong University (Other)
Responsible Party: Principal Investigator, Yanqing Li, Vice President, Chief of the Department of Gastroenterology, Qilu Hospital, Shandong University, Shandong University
Other Study IDs: 2012SDU-QILU-G01
Record Dates: First submitted 2012-06-28; First posted 2012-07-20 (Estimated); Last update posted 2012-07-20 (Estimated); Status verified 2012-07

CONDITIONS: Gastric Intestinal Metaplasia
Keywords: Gastric Intestinal Metaplasia; Confocal Laser Endomicroscopy

STUDY DESIGN:
Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Taken biopsies during endoscopy
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- Consecutive patients for CLE examination
  Interventions: Procedure: CLE examination for upper gastrointestinal tract

INTERVENTIONS:
Procedure: CLE examination for upper gastrointestinal tract — Routine upper GI endoscopy plus targeted CLE examination
  Other Names: confocal endomicroscopy

SUMMARY:
The study aims to:

1. Explore the properties of mesenchymal black spots, and to determine the value of mesenchymal black spots in diagnosing gastric intestinal metaplasia by confocal laser endomicroscopy (CLE).
2. Evaluate the incidences of gastric intraepithelial neoplasia and gastric cancer in patients with gastric mesenchymal black spot during CLE imaging.

DETAILED DESCRIPTION:
Gastric intestinal metaplasia (GIM) is confirmed to be a risk factor that may lead to the development of intestinal type gastric cancer. Previous study has shown that confocal laser endomicroscopy promising in the diagnosis of GIM. The investigators have found an elevated incidence of mesenchymal black spots in patients with GIM during previous CLE imaging. This study aims to explore the properties of mesenchymal black spots, and to determine the value of mesenchymal black spots in diagnosing gastric intestinal metaplasia by confocal laser endomicroscopy.

ELIGIBILITY:
Inclusion Criteria:

* Patients will include male or female aged between 18 and 80 years with indications for upper-endoscopy , but without any disease of heart, liver or kidney.

Exclusion Criteria:

* Patients who are allergic to fluorescein sodium
* Patients who are unwilling to sign or give the informed consent form
* Patients with impaired cardiac, liver or renal function
* Patients with coagulopathy
* Patients with pregnancy or breastfeeding

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients without any disease of heart, liver or kidney.
Sampling Method: Non-Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2012-06; Primary Completion 2012-12 (Estimated); Study Completion 2012-12 (Estimated)

PRIMARY OUTCOMES:
Accuracy of black spots in diagnosis of gastric intestinal metaplasia | up to six months

CONTACTS AND LOCATIONS:
Overall Officials: Yanqing Li, MD, PhD, Study Director — Department of Gastroenterology, Qilu Hospital
Locations (1):
- Department of Gastroenterology, Qilu Hospital, Shandong University, Jinan, Shandong, China